CLINICAL TRIAL: NCT04674943
Title: Effects of Breathing Exercises on Asthmatic Pregnant Females
Brief Title: Breathing Exercises in Asthma During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00702 Saba Seemab
Record Dates: First submitted 2020-12-16; First posted 2020-12-19 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Asthma in Pregnancy
Keywords: Asthma; Forced Expiratory volume in 1 sec (FEV1); Forced Vital capacity (FVC); Peak Expiratory flow rate; Pregnancy; Quality of life
MeSH Terms: conditions — Asthma | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No physical therapy intervention was given. Only pharmacological treatment was provided.
- Breathing exercise group (Experimental): 1. Pursed lip breathing 15 reps x 3 sets) 2: Diaphragmatic breathing (15 reps x 3 sets) 3:Lateral costal breathing 15 reps x 3 sets)
  Interventions: Other: Breathing exercises

INTERVENTIONS:
Other: Breathing exercises — Breathing exercises as well as Buteyko technique and Papworth relaxation method was performed as relaxation technique. All exercises were performed 15rep 3 sets for 15 min.
  Arms: Breathing exercise group

SUMMARY:
The aim of this research is to determine the effects of breathing exercises on asthmatic pregnant females. A randomized controlled trial will be done for which the calculated sample size is 24. Non probability purposive sampling technique will be used and the subjects will be randomly divided in two groups, with one group undergoing pharmacological management where as breathing exercises will be provided to the other group. Lung volumes and capacities as well as quality of life will be assessed through questionnaire in order to determine the effect of breathing exercises in patients with asthma.

DETAILED DESCRIPTION:
Asthma is defined as chronic inflammatory condition of airways, characterized by periodic episodes of wheezing, cough, chest tightness, shortness of breath and which are often worse at night. This causes hyper-responsiveness of airways and flow of air obstruction leading to breathing difficulty. Asthma in pregnancy is a common risk factor for fetal and maternal complications. Asthma also effects outcomes of pregnancy and pregnancy affects asthma severity which has being currently being examined.

Approximately 50% of asthmatic pregnant females 25 percent experience a worsening of asthma control at some stage during pregnancy, and most of them take corticosteroids for the management of acute and chronic exacerbation. Pathogenesis of asthma during pregnancy is entirely related to the physiological and pathological changes .Uterine enlargement causes hormonal changes during pregnancy directly or indirectly Asthmatic women have an increased ratio of associated co-morbidities which have direct effect on it where by increasing risk of perinatal outcomes. Pregnancy associated with asthma affects women in many ways. Hormonal imbalances occurring during pregnancy affects lungs as well as sinuses. Increased estrogen causes nasal congestion during the 3rd trimester. A rise in progesterone may cause a feeling of shortness of breath. Its important to identify or diagnose asthma being a major cause of shortness of breath during pregnancy. Breathing exercises includes nasal breathing, diaphragmatic breathing, deep pursed lip breathing. They have beneficial effects, such as betterment in health related (QOL)quality of life ,decreasing anxiety ,depression, improving asthma symptoms, the treatment using relief medication, occurrence of exacerbations, and hyperresponsiveness of airways.

Global Initiative for Asthma(GINA GUIDELINES 2019)illustrated that non pharmacological management such as patient's education, breathing exercises and relaxation techniques can be used as an adjunct to asthma pharmacotherapy. Breathing exercises includes nasal breathing, diaphragmatic breathing, deep pursed lip breathing. They have beneficial effects, such as betterment in health related (QOL)quality of life, decreasing anxiety ,depression, improving asthma symptoms, the treatment using relief medication, occurrence of exacerbations, and hyperresponsiveness of airways in patients with asthma. Literature reviewed from different search engines shows that there are limited studies available regarding non pharmacological management of asthma during pregnancy so Current study is planned to assess if non pharmacological management such as breathing exercise techniques will help improve asthma symptoms exacerbation as well as quality of life following regular plan of exercises and relaxation techniques collectively.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 20-40years
* Gestational week 13 to 28 weeks
* Asthma in women with mild and intermittent asthma
* Asthma in women with active mild and persistent asthma

Exclusion Criteria:

* Patents with any psychological disorder
* Patients with neurological, musculoskeletal, cardiac and pulmonary disease and physical impairments

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Study is going to be conducted on female pregnant patients with asthma
Enrollment: 24 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate (PEFR) | 4 weeks
  Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.
Forced vital capacity (FVC) | 4 weeks
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
Forced expiratory volume in 1sec (FEV1) | 4 weeks
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
FVC/FEV1 | 4 weeks
  FVC/FEV1 measured through digital spirometer. The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65).
Asthma Control Questionnaire | 4 weeks
  Asthma Control questionnaire is a self-reported subjective outcome measurement tool that is used to measure the sufficiency of asthma symptom control and changes in asthma symptoms. It is 5 point scale with scores ranging from 0 to 5 for each item. The greater the score of Asthma Control questionnaire, the better the prognosis and outcome.

SECONDARY OUTCOMES:
Quality of life questionnaire (Short form 36) - SF 36 | 4 weeks
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health which indicates quality of life with regard to different health domains.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy VE, Gibson PG. Asthma in pregnancy. Clin Chest Med. 2011 Mar;32(1):93-110. doi: 10.1016/j.ccm.2010.10.001. Epub 2010 Dec 17. PMID 21277452
- [Background] Wang H, Li N, Huang H. Asthma in Pregnancy: Pathophysiology, Diagnosis, Whole-Course Management, and Medication Safety. Can Respir J. 2020 Feb 22;2020:9046842. doi: 10.1155/2020/9046842. eCollection 2020. PMID 32184907
- [Background] Murphy VE. Managing asthma in pregnancy. Breathe (Sheff). 2015 Dec;11(4):258-67. doi: 10.1183/20734735.007915. PMID 27066119
- [Background] Tan KS, Thomson NC. Asthma in pregnancy. Am J Med. 2000 Dec 15;109(9):727-33. doi: 10.1016/s0002-9343(00)00615-x. PMID 11137489
- [Background] Labor S, Dalbello Tir AM, Plavec D, Juric I, Roglic M, Pavkov Vukelic J, Labor M. What is safe enough - asthma in pregnancy - a review of current literature and recommendations. Asthma Res Pract. 2018 Dec 27;4:11. doi: 10.1186/s40733-018-0046-5. eCollection 2018. PMID 30607253
- [Background] Evaristo KB, Mendes FAR, Saccomani MG, Cukier A, Carvalho-Pinto RM, Rodrigues MR, Santaella DF, Saraiva-Romanholo BM, Martins MA, Carvalho CRF. Effects of Aerobic Training Versus Breathing Exercises on Asthma Control: A Randomized Trial. J Allergy Clin Immunol Pract. 2020 Oct;8(9):2989-2996.e4. doi: 10.1016/j.jaip.2020.06.042. Epub 2020 Aug 6. PMID 32773365